CLINICAL TRIAL: NCT03497897
Title: A Randomized, Subject and Investigator Blinded, Placebo Controlled, Multi-center Study in Parallel Groups to Assess the Efficacy and Safety of LYS006 in Patients With Moderate to Severe Inflammatory Acne
Brief Title: Study to Assess the Efficacy and Safety of LYS006 in Patients With Moderate to Severe Inflammatory Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLYS006X2201; 2017-003191-30 (EudraCT Number)
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Inflammatory Acne
Keywords: Acne, efficacy, safety
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LYS006 20 mg BID (Experimental): LYS006, 20 mg, orally, twice daily (BID), for 12 weeks
  Interventions: Drug: LYS006 20 mg
- LYS006 2 mg BID (Experimental): LYS006, 2 mg, orally, BID, for 12 weeks
  Interventions: Drug: LYS006 2 mg
- Placebo BID (Placebo Comparator): Matching placebo, orally, BID, for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LYS006 20 mg — LYS006 20 mg, capsules, oral administration, BID, for 12 weeks
  Arms: LYS006 20 mg BID
Drug: LYS006 2 mg — LYS006 2 mg, capsules, oral administration, BID, for 12 weeks
  Arms: LYS006 2 mg BID
Drug: Placebo — Matching placebo, capsules, oral administration, BID, for 12 weeks
  Arms: Placebo BID

SUMMARY:
The main purpose of this study is to assess preliminary efficacy and safety of LYS006 in patients with moderate to severe inflammatory acne and to determine if LYS006 has an adequate clinical profile for further clinical development.

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, subject- and investigator-blinded, multicenter, nonconfirmatory, parallel group, and proof-of-concept study in adult patients with moderate to severe inflammatory acne. After an initial screening period (up to 4 weeks), subjects were treated with LYS006 or matching placebo for 12 consecutive weeks to assess preliminary clinical efficacy, safety, and tolerability in the targeted subject population. At the beginning of the treatment period, subjects were randomized to one of three treatment groups, i.e., LYS006 20 mg twice daily (BID), LYS006 2 mg BID or matching placebo in a 3:1:3 ratio.

After treatment period completion, all subjects entered a post-treatment safety follow-up period of 4 weeks without study drug administration. The maximum duration of study participation was 20 weeks. Study completion was defined as when the last subject completed his/her study completion visit, and any repeat assessments associated with this visit were documented and followed-up appropriately by the investigator, or in the event of an early study termination decision, the date of that decision.

ELIGIBILITY:
Inclusion criteria:

* Male and female subjects aged 18 to 45 years of age inclusive, and otherwise in good health as determined by medical history, physical examination, vital signs, ECGs and laboratory tests at screening.
* Body weight between 50 and 120 kg, both inclusive, at screening.
* Patients with papulo-pustular acne vulgaris (inflammatory acne) presenting with 20 to 100 facial inflammatory lesions (papules, pustules and nodules) at baseline, no more than 2 facial inflammatory nodules or cysts at screening and baseline, and a minimun number of 10 non-inflammatory facial lesions (open and closed comedones).
* Patients who are candidates for systemic treatment and for whom in the opinion of the investigator, an appropriate previous treatment with topical anti-acne medication failed, or was not well tolerated, or is not indicated (e.g., due to large body surface area affected, e.g., on the back)
* Patients with Grade 3 (moderate) or Grade 4 (severe) IGA score assessed by the investigator at screening and baseline.

Exclusion criteria:

* Appropriate wash out periods are required for investigational drugs, any oral/systemic treatment for acne, systemic or lesional injected (for acne) corticosteroids or systemic immunomodulators, any systemic hormonal treatments, previous treatment with biologics, oral retinoids (in particular isotretinoin) and any topical anti-acne treatment.
* Previous surgical, physical (such as ThermaClear™), light (including blue or UV light, photodynamic therapy or laser therapy within 4 weeks prior to baseline
* Use of facial medium depth chemical peels (excluding home regimens) within 3 months prior to baseline.
* Any other forms of acne
* Any severe, progressive or uncontrolled medical or psychiatric condition or other factors at randomization that in the judgment of the investigator prevents the patient from participating in the study.
* Active systemic infections (other than common cold) during the 2 weeks prior to baseline.
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result at screening.
* Chronic infection with Hepatitis B or Hepatitis C virus.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive Human chorionic gonadotropin (HCG) laboratory test.
* Sexually active males or women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of study treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (7):
  - Novartis Investigative Site, Fremont, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Hialeah, Florida
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Pflugerville, Texas
- Novartis Investigative Site, Pilsen, Czechia
- Novartis Investigative Site, Nice, France
- Germany (4):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Frankfurt
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — http://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 18 investigative sites in 6 countries.
Pre-assignment Details: There was an initial screening period of up to 4 weeks.
Period: Overall Study
Arm/Group | LYS006 20 mg BID | LYS006 2 mg BID | Placebo BID
Started | 26 | 11 | 29
Completed Treatment Period | 23 | 9 | 24
Pharmacodynamic (PD) Analysis Set (The PD analysis set included all participants with available PD data who received any study drug and with no protocol deviations with relevant impact on PD data.) | 24 | 11 | 28
Completed (Participants who completed the study) | 20 | 9 | 23
Not Completed | 6 | 2 | 6
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Subject/Guardian Decision | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LYS006 20 mg BID | LYS006 2 mg BID | Placebo BID | Total
Number analyzed (Participants) | 26 | 11 | 29 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (6.89) | 24.5 (6.23) | 25.0 (5.40) | 24.2 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 22 | 46
  Male | 10 | 3 | 7 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 1 | 3
  Black or African American | 2 | 1 | 6 | 9
  Other | 2 | 1 | 6 | 9
  White | 21 | 8 | 16 | 45

OUTCOME MEASURES:

1. Primary Outcome: Total Inflammatory Lesion Count
Description: Inflammatory facial lesion count included papules, pustules, and nodules. The natural log transformed inflammatory facial lesion count up to Week 12 was analyzed using a Bayesian mixed effect model for repeated measurements (MMRM). Values estimated from the model at Week 12 are presented in the table. Posterior geometric mean and 90% credible intervals in each group are presented.
Time Frame: Week 12
Population: Participants in the PD analysis set who had a valid assessment of the outcome measure.
Measure: Geometric Mean (90% Confidence Interval); unit: lesions
Arm/Group | LYS006 20 mg BID | LYS006 2 mg BID | Placebo BID
Number analyzed (Participants) | 21 | 9 | 23
lesions | 18.55 [14.16 to 24.32] | 24.51 [16.35 to 36.94] | 20.04 [15.42 to 26.13]
Statistical Analysis 1: Comparison: LYS006 20 mg BID vs Placebo BID; Test type: Other — The effects included in the model are: log transformed baseline inflammatory facial lesion count, treatment group, visit, treatment group by visit interaction, log transformed baseline inflammatory facial lesion count by visit interaction and type of center; Bayesian analysis; Bayesian mixed effect model with repeated measures; Posterior geometric mean ratio = 0.93, 90% CI 2-sided [0.64 to 1.34] — 90% credible intervals are reported on the geometric means ratio
Statistical Analysis 2: Comparison: LYS006 20 mg BID vs Placebo BID; Test type: Other — [test comment as in outcome 1, analysis 1]; Bayesian analysis; Bayesian mixed effect model with repeated measures; P(Geometric Mean Ratio<1) = 0.637 — Posterior probability on geometric mean ratio is reported
Statistical Analysis 3: Comparison: LYS006 20 mg BID vs Placebo BID; Test type: Other — [test comment as in outcome 1, analysis 1]; Bayesian analysis; Bayesian mixed effect model with repeated measures; P(Geometric Mean Ratio<0.75) = 0.171 — Posterior probability on geometric mean ratio is reported

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 128 days
Groups:
- Total: Total
Arm/Group | LYS006 20 mg BID | LYS006 2 mg BID | Placebo BID | Total
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/11 | 0/29 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/11 | 0/29 | 0/66
Other Adverse Events (participants affected / at risk) | 10/26 | 8/11 | 16/29 | 34/66
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LYS006 20 mg BID (N=26) | LYS006 2 mg BID (N=11) | Placebo BID (N=29) | Total (N=66)
Haemoglobinaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Fatigue (General disorders) | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 1
Genital infection fungal (Infections and infestations) | 1 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3 | 3 | 9
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Urethritis (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 4
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Albumin urine present (Investigations) | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Bacterial test positive (Investigations) | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 3 | 6
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Blood urine present (Investigations) | 1 | 0 | 0 | 1
Creatinine urine increased (Investigations) | 1 | 0 | 0 | 1
Crystal urine present (Investigations) | 2 | 0 | 4 | 6
Haematocrit increased (Investigations) | 1 | 0 | 1 | 2
Haemoglobin increased (Investigations) | 0 | 0 | 2 | 2
Lipase increased (Investigations) | 0 | 0 | 1 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 1
Protein urine present (Investigations) | 1 | 0 | 1 | 2
Urine protein/creatinine ratio increased (Investigations) | 2 | 1 | 1 | 4
White blood cell count increased (Investigations) | 0 | 0 | 1 | 1
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 3 | 5
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria aquagenic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT03497897/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT03497897/SAP_001.pdf